CLINICAL TRIAL: NCT00643019
Title: Preventing Recurrent Sexually Transmitted Infections in Minority Women
Brief Title: Project Sexual Awareness for Everyone (SAFE)
Acronym: SAFE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC2004415H; U01AI040029 (NIH)
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Sexually Transmitted Disease; Secondary Prevention; Behavioral Modification; Public Health
Keywords: Sexually Transmitted Infections; Secondary Prevention; Cognitive Behavioral Intervention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SAFE Intervention (Experimental): Behavioral Intervention
  Interventions: Behavioral: SAFE Behavioral Intervention
- Control (Other): Sexually Transmitted Infection Risk Reduction Counseling
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: SAFE Behavioral Intervention — Group cognitive behavioral intervention sessions
  Arms: SAFE Intervention
Other: Control — Individual Sexually Transmitted Infection Risk Reduction Counseling
  Arms: Control

SUMMARY:
This trial randomizes young Mexican American and African American women with a sexually transmitted infection to a behavioral intervention (3 three hour weekly sessions) versus control with the goal of preventing recurrent sexually transmitted infections.

DETAILED DESCRIPTION:
Participants are interviewed, examined, and offered treatment at 0, 6, 12 months and as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Mexican American,
* 14 - 45 years old,
* English Speaking,
* non-viral sexually transmitted infection

Exclusion Criteria:

* Non-English speaking,
* viral sexually transmitted infection

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 800 (Estimated)
Dates: Start 1993-01; Primary Completion 1994-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Re-infection with a non-viral sexually transmitted infection | 1 year

SECONDARY OUTCOMES:
Changes in risky sexual behavior | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle N Shain, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Sciences Center San Antonio, San Antonio, Texas, United States

REFERENCES:
- [Derived] Thurman AR, Holden AE, Shain RN, Perdue S, Piper JM. Preventing recurrent sexually transmitted diseases in minority adolescents: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1417-25. doi: 10.1097/AOG.0b013e318177143a. PMID 18515527